CLINICAL TRIAL: NCT03031678
Title: Office of Device Evaluation Lead-MED-EL EAS Extended f/u Study
Brief Title: Electric-Acoustic Stimulation Extended Follow-up Post Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P000025/PAS001
Record Dates: First submitted 2017-01-13; First posted 2017-01-25 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study procedures (Other)
  Interventions: Device: Electric-Acoustic Stimulation (EAS) Cochlear Implant System

INTERVENTIONS:
Device: Electric-Acoustic Stimulation (EAS) Cochlear Implant System — Combination of a cochlear implant and a hearing aid
  Other Names: EAS

SUMMARY:
The MED-EL EAS Extended Follow-up Study is an extended follow-up of the subjects who were enrolled in the pivotal study to assess long-term safety and device performance.

DETAILED DESCRIPTION:
The study will be conducted as a prospective, non-controlled, non-randomized, multicenter study at the 14 sites. Up to 68 available subjects who were enrolled in the pivotal study will be invited to participate in the extended follow-up. Study subjects will be followed for a minimum of 5 years post-implantation of the device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of implantation
* Severe to profound sensorineural hearing loss for frequencies greater than 1500 Hz (i.e., threshold no better than 70 dB HL at 2000-8000 Hz)
* Low-frequency thresholds up to and including 500 Hz no poorer than 65 dB HL
* CNC word recognition score less than or equal to 60% in the ear to be implanted
* CNC word recognition score less than or equal to 60% in the contralateral ear
* English spoken as the primary language

Exclusion Criteria:

* Conductive, retrocochlear, or central auditory disorder
* Hearing loss in the ear to be implanted that has demonstrated a recent fluctuation at two or more frequencies of 15 dB in either direction in the last 2 years
* Any physical, psychological, or emotional disorder that interferes with surgery or the ability to perform on test and rehabilitation procedures
* Developmental delays or organic brain dysfunction
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations
* Unwillingness or inability of the candidate to comply with all investigational requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford Unversity, Palo Alto, California
  - University of Miami, Miami, Florida
  - University of Kansas University Medical Center, Kansas City, Kansas
  - University of North Carolina, Chapel Hill, North Carolina
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Skarzynski H, van de Heyning P, Agrawal S, Arauz SL, Atlas M, Baumgartner W, Caversaccio M, de Bodt M, Gavilan J, Godey B, Green K, Gstoettner W, Hagen R, Han DM, Kameswaran M, Karltorp E, Kompis M, Kuzovkov V, Lassaletta L, Levevre F, Li Y, Manikoth M, Martin J, Mlynski R, Mueller J, O'Driscoll M, Parnes L, Prentiss S, Pulibalathingal S, Raine CH, Rajan G, Rajeswaran R, Rivas JA, Rivas A, Skarzynski PH, Sprinzl G, Staecker H, Stephan K, Usami S, Yanov Y, Zernotti ME, Zimmermann K, Lorens A, Mertens G. Towards a consensus on a hearing preservation classification system. Acta Otolaryngol Suppl. 2013;(564):3-13. doi: 10.3109/00016489.2013.869059. PMID 24328756

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Procedures
Started | 50
EAS Test Condition Complete | 39
CI Alone Test Condition Complete | 10
Completed | 49
Not Completed | 1
Not completed — Study closed prior to completion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Procedures
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.58 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50
Ear Implanted [Count of Participants; unit: Participants]
  Right | 27
  Left | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Words Correct As Assessed by CUNY Sentence Test.
Description: Long-term effectiveness of the Electric-Acoustic System will be assessed by speech perception testing in noise with CUNY sentences completed through five years post-implantation.
Time Frame: Five years (60 months) post-implantation for subjects implanted under the original EAS clinical trial
Measure: Mean (Standard Deviation); unit: percentage of words correct
Groups:
- Electric Acoustic Stimulation: Subjects tested with a combination of electric and acoustic stimulation
- CI Alone: Subjects testing with electric stimulation only
Arm/Group | Electric Acoustic Stimulation | CI Alone
Number analyzed (Participants) | 39 | 10
percentage of words correct | 61.33 (27.05) | 43.30 (33.10)

2. Secondary Outcome: Classification of Residual Hearing at 5 Years Post Operatively as a Function of the HEARRING SCALE.
Description: The HEARRING Scale was developed by the HEARRING Research Group, a collaboration of surgeons and audiologists in the hearing implant field who work together to develop consensus statements. The Scale was published in 2013 by Skarzynski et al. as means to classify post-operative residual hearing thresholds. Residual hearing is classified as complete (100-76%), partial (26-75%), minimal (1-25%), or none (0%) according to an equation which takes into account pre-operative thresholds, post-operative thresholds, and the limits of the audiometer.
Time Frame: Five years (60 months) post-implantation for subjects implanted under the original EAS clinical trial
Measure: Count of Participants; unit: Participants
Arm/Group | Study Procedures
Number analyzed (Participants) | 50
Participants
  Complete Hearing Preservation | 6
  Partial Hearing Preservation | 31
  Minimal Hearing Perservation | 9
  No Hearing Preservation | 4

3. Secondary Outcome: Percentage of Words Correct as Assessed by CNC Words in Quiet.
Description: Long-term effectiveness of the Electric-Acoustic System will be assessed by speech perception testing in quiet with CNC words completed through five years post-implantation.
Time Frame: Five years (60 months) post-implantation for subjects implanted under the original EAS clinical trial
Measure: Mean (Standard Deviation); unit: percentage of words correct
Groups:
- Electric Acoustic Stimulation: Subjects tested with electric and acoustic stimulation combined
- CI Alone: Subjects tested with electric stimulation only
Arm/Group | Electric Acoustic Stimulation | CI Alone
Number analyzed (Participants) | 39 | 10
percentage of words correct | 73.59 (13.71) | 57.40 (23.29)

4. Secondary Outcome: Subjective Benefit From EAS Through 5 Years Post Implantation Measured on the APHAB (Abbreviated Profile Hearing Aid Benefit) Questionnaire.
Description: The APHAB Questionnaire measures percentage of listening difficulty on a scale from 100% (very difficult) to 0% (not difficult at all). Results are reported as the average listening difficulty across subjects.
Time Frame: Five years (60 months) post-implantation for subjects implanted under the original EAS clinical trial
Population: 46 completed the questionnaire
Measure: Mean (Standard Deviation); unit: percentage of listening difficulty
Arm/Group | Study Procedures
Number analyzed (Participants) | 46
percentage of listening difficulty | 35.39 (13.89)

ADVERSE EVENTS:
Time Frame: 3 Years (Duration of the Study)
Description: Any adverse event reported by a subject over the duration of the study is included here. Subjects were monitored through at least five years post-implantation from the original clinical trial.
Arm/Group | Study Procedures
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Procedures (N=50)
Loss of Residual Hearing (Ear and labyrinth disorders) | 7 (7)
Internal Device Failure (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03031678/Prot_SAP_000.pdf